# All in Dads! Healthy Marriage and Responsible Fatherhood Program Evaluation

Study Protocol

NCT05194020

October 17, 2024

The purpose of this information collection is to document local evaluation plans conducted as part of the *Fatherhood Family-Focused, Interconnected, Resilient, and Essential (Fatherhood FIRE)* grants. Public reporting burden for this collection of information is estimated to average 8 hours per response, including the time for reviewing instructions, gathering and maintaining the data needed, and reviewing the collection of information. This is a voluntary collection of information. An agency may not conduct or sponsor, and a person is not required to respond to, a collection of information subject to the requirements of the Paperwork Reduction Act of 1995, unless it displays a currently valid OMB control number. The OMB # is 0970-0356 and the expiration date is 06/30/2021. If you have any comments on this collection of information, please contact Charles Michalopoulos@mdrc.org.

## **FATHERHOOD FIRE EVALUATION PLAN**

# **GLOSSARY OF TERMS**

There are different types of program evaluations and many different ways to describe them. To facilitate communication, the terms used here are described below:

- Implementation Evaluation: An evaluation that addresses the extent to which a
  program is operating as intended. It describes who participated in the program, the
  services they received, and how services were provided. It assesses program operations
  and whether the population targeted was served. Implementation evaluation helps
  identify why a program's intended outcomes were or were not achieved. Implementation
  evaluation cannot address whether changes have occurred as a result of the program. It
  is also called a process evaluation or formative evaluation.
- Outcome Evaluation: Outcome evaluation is used to measure the results of a program.
  It assesses whether the program led to intended changes in participants' knowledge, skills, attitudes, behaviors, or awareness. It can be descriptive or impact depending on whether it seeks to address whether the intended changes were the result of the program.
- Impact Evaluation: Impact evaluation is a type of outcome evaluation that attributes participant changes to the program. To do so, it includes a comparison or control group to help establish that program activities, not something else, caused the changes in the observed outcomes. In this design, two groups are included in the evaluation: (1) a treatment group that includes individuals who participate in the program; and (2) a comparison group that includes individuals who are similar to those in the treatment group, but who do not receive the same services.
- Descriptive Evaluation: Descriptive evaluation is a type of outcome evaluation that measures change in outcomes by making comparisons among participants after

program participation and conditions prior to participation. This design involves collecting information only on individuals participating in the program. This information is collected at least twice: once before participants begin the program and sometime after they complete program.

## PROGRAM BACKGROUND

## 1. PROGRAM SUMMARY

Please provide a brief summary of your grant project including the needs to be addressed, the services provided, and the population served.

The purpose of this project is to help fathers establish and strengthen their relationship with their children and the mothers of their children; to reduce domestic violence in vulnerable families; to improve economic stability of fathers through comprehensive, job-driven career services; to employ intensive case management barrier removal, individual job coaching, and comprehensive family development to improve short and long-term outcomes.

The target population for this project are low-income urban father in high poverty and high-risk neighborhoods who are above the age of 18 with children under the age of 24. These fathers include non-custodial and custodial fathers, TANF eligible fathers, fathers at or below federal poverty levels, and fathers with children in early childhood learning centers. This project also focuses on fathers who have been or may be at risk of domestic violence (victims and perpetrators), under-involved or uninvolved in their children's lives, unemployed, underemployed, lacking in education (GED/diploma), in need of job skills, or experiencing the following barriers: criminal records, mental health conditions, addictions, or disabilities.

This project is needed in this community because Franklin County is the most populous county in Ohio with 1.3 million residents and a poverty rate of 16.7%. The largest city in Franklin County, Columbus, has a poverty rate of 20.2% for all residents but 31.4% among black residents and 32.1% among Hispanic residents. Furthermore, in the seven Columbus zip codes targeted in this project, the average poverty rate is 45.1%. The Columbus Metro region is one of the most racially and economically segregated regions in the country.

This persistent and pervasive poverty negatively impacts upward mobility of families, exacerbates disparities, and reinforces generational poverty. Additionally, in Ohio, 1 in 3 women and 1 in 4 men have experienced some form of physical violence by an intimate partner which accounts for 15% of all violent crime. Since March 2020 there has been a 20% increase in domestic violence calls due to COVID-19 shutdowns and US Labor Department data shows the national unemployment rate among blacks has tripled. Funds from this grant will be used to address, support, and integrate all three authorized activities: Responsible Fatherhood, Healthy Marriage and Relationships, and Economic Stability.

All In Dads! will take an integrated and comprehensive approach utilizing parenting education, intensive case management, coaching, mentoring, and employment services to improve long-term outcomes for our target population. All In Dads! will educate fathers and couples to improve the quality of and increase the frequency of father/child engagement, improve spousal/co-parent-parenting pair relationships, reduce conflict and domestic violence, and create safer and happier families by improving child and parent well-being, self-esteem, and health.

#### 2. EVALUATION GOALS

Please briefly describe key goals of your evaluation and what you hope to learn below.

The goals for the AFC Fatherhood project are improved family functioning (parenting and coparenting), improved adult and child well-being, increased economic stability and mobility, and reduced poverty by providing intensive, integrated services in promoting responsible parenting and economic stability with funds from The Fatherhood Family-Focused Interconnected, Resilient and Essential Grants. Evaluation goals include achieving sufficient sample size, retaining participants through the use of incentives, collecting valid and complete data, and ultimately making a contribution to the field of responsible fatherhood in the literature.

## 3. EVALUATION ENROLLMENT

Please provide the expected start and end dates for program and evaluation enrollment using the tables below. For impact studies, please indicate expected start and end dates for each study group.

| <b>DESCRIPTIVE EVALUATION</b> Please leave blank if not conducting a descriptive outcome evaluation. | | |
|---|---|---|
| Program Enrollment Study Enrollment | | |
| Start Date | 4/1/2021 | 4/1/2021 |
| End Date | 9/30/2025 | 3/31/2024 |
| Definition | All participants enrolled for services | All participants enrolled for services to include local evaluation |

# 4. EVALUATION TIMELINE

Please include a timeline for key activities of the evaluation below. Example of activities may include IRB submission, staff training, waves of data collection, analysis period, and report writing and submission.

| Evaluation Activity | Start Date | End Date |
|---|---|---|
| Additional Evaluation staff hiring and onboarding | 1/15/2021 | 2/15/2021 |
| Evaluation staff training | 1/22/2021 | 2/20/2021 |
| Evaluation Kickoff meeting and orientation with all program staff | 2/2/2021 | 2/3/2021 |
| IRB training and certification by all program and evaluation staff | 10/1/2020 | 2/28/2021 |
| Development and submission of Evaluation Plan document | 1/15/2021 | 2/19/2021 |
| Evaluation Tools Development | 10/1/2020 | 2/28/2021 |
| IRB Approval | 3/1/2021 | 3/15/2021 |
| CQI Team Formed and Meeting bi-weekly | 3/15/2021 | 7/1/2025 |
| Training for CQI Team | 3/15/2021 | 3/28/2021 |
| Training for all Program Staff on Research Methods and process | 3/15/2021 | 3/28/2021<br>+ Refreshers as<br>needed including new<br>staff |
| Evaluation Data Collection | 4/1/2021 | 5/31/2025 |
| Baseline Data | 4/1/2021 | 3/31/2024 |
| Post Test Data | 5/17/2021 | 8/2/2024 |
| Follow-up Data | 4/1/2022 | 5/31/2025<br>at the latest |
| 1 <sup>st</sup> Manuscript submitted for publication | 7/1/2025 | 12/31/2025 |

# **EVALUATION PLAN**

## 1. RESEARCH QUESTIONS

## 1.1. OVERVIEW OF RESEARCH QUESTIONS

Please state the research questions(s) that the evaluation intends to answer and for each research question indicate the type: implementation or outcome.

- Implementation Questions: Identifying whether a program has been successful in attaining desired implementation goals (e.g., reaching intended target population, enrolling intended number of participants, delivering training and services in manner intended, etc.)
- Outcome Questions: Identifying whether program is associated with intended outcomes for participants (e.g., do participants' knowledge, attitudes, behaviors, or awareness change?)

Research questions in this study are framed by a Descriptive Evaluation Design to assess whether outcomes improve for low-income fathers who participate in the All in Dads! (AID!) Project. Primary and secondary outcomes are assessed before and after participants complete core curricula—Father Factor, The New Playbook, and Money Smart—and Job Readiness Coaching and Career Development as employment support services (pre to post). Primary outcome measures will indicate whether behavior improved for healthy family relationships (parent, co-parent, and partner). Secondary outcome measures will indicate whether behavior improved for the attitudes and expectations that facilitate and reflect behavior for healthy family relationships and economic stability (financial, employment) (see Table 1 below).

| No | Research Question | Implementation or Outcome? |
|---|---|---|
| R1 | Will participants report significantly <b>healthier parenting behavior</b> one-year after completing primary educational services and employment support services? | Primary Outcome |
| R2 | Will participants report significantly <b>healthier co-parenting behavior</b> one-year after completing primary educational services and employment support services? | Primary Outcome |
| R3 | Will participants report significantly <b>healthier financial behavior</b> one-year after completing primary educational services and employment support services? | Secondary Outcome |
| R4 | Will participants report significantly <b>healthier parenting attitudes</b> after completing primary educational services and employment support services? | Secondary Outcome |

# 1.2. OUTCOME RESEARCH QUESTIONS

For each <u>outcome research question</u> listed above, whether a descriptive or impact design, summarize the inputs (e.g., program components, program supports, implementation features, etc.), target population (e.g., the population for which the effect will be estimated) and the outcomes (e.g., child well-being, father-child engagement, etc.) that will be examined to answer the research question(s). Comparisons for descriptive evaluations may reflect circumstances before the grant, pre-treatment, or pre-determined benchmark from other studies with similar interventions.

| Research<br>Question<br>Number<br>Should<br>correspond<br>to the<br>number<br>indicated<br>in Table<br>1.1 above | Intervention Program component or set of activities that the evaluation will test or examine | Target Population Population for which the effect of the treatment will be estimated | Comparison What the intervention will be compared to (e.g., pre-intervention for descriptive designs) | Outcome Changes that are expected to occur as a result of the intervention | Confirmatory or Exploratory? Confirmatory: those upon which conclusions will be drawn Exploratory: those that may provide additional suggestive evidence |
|---|---|---|---|---|---|
| R1 | Primary curricula (Father Factor, The New Playbook, and Money Smart); Employment Support (Job Readiness Coaching, Career Development); Continuous Quality Improvement (CQI) Process | Low-income fathers who are 18+ years with children up to 24 years who are residents of Franklin County in Ohio | Assessment of healthy parenting behavior at AID! Project enrollment. | Participants who complete primary and support services will report healthier parenting behavior one year after AID! enrollment. | Confirmatory |
| R2 | Primary curricula (Father Factor, The New Playbook, and Money Smart); Employment Support (Job Readiness Coaching, Career Development); | Low-income fathers who are 18+ years with children up to 24 years who are residents of Franklin County in Ohio | Assessment of healthy coparenting behavior at AID! Project enrollment. | Participants who complete primary and support services will report healthier coparenting behavior one year | Confirmatory |

| | Continuous<br>Quality<br>Improvement<br>(CQI) Process | | | after AID! enrollment. | |
|---|---|---|---|---|---|
| R3 | Primary curricula (Father Factor, The New Playbook, and Money Smart); Employment Support (Job Readiness Coaching, Career Development); Continuous Quality Improvement (CQI) Process | Low-income fathers who are 18+ years with children up to 24 years who are residents of Franklin County in Ohio | Assessment of healthy financial behavior at AID! Project enrollment. | Participants who complete primary and support services will report healthier financial behavior one year after AID! enrollment. | Confirmatory |
| R4 | Primary curricula (Father Factor, The New Playbook, and Money Smart); Employment Support (Job Readiness Coaching, Career Development); Continuous Quality Improvement (CQI) Process | Low-income fathers who are 18+ years with children up to 24 years who are residents of Franklin County in Ohio | Assessment of healthy parenting attitudes immediately following program completion post-intervention. | Participants who complete primary and support services will report healthier parenting attitudes immediately following program completion | Confirmatory |

# 2. BACKGROUND

For each <u>outcome research question listed in 1.1</u>, whether descriptive or impact design, briefly summarize the previous literature or existing research that informs the stated research question and how the evaluation will expand the evidence base. Explain why the research questions are of specific interest to the program and/or community. Only a short summary paragraph

description is needed below. Additional documentation, such as a literature review, may be appended to this document.

| Research<br>Question | Existing Research | Contribution to the Evidence Base | Interest to the Program and/or Community |
|---|---|---|---|
| R1 | Low-income fathers can lack the <b>parenting skills</b> to fulfill their familial obligations as a parent to promote healthy family relationships. | Determine the extent to which the delivery of AID! Project services enhance the parenting skills of low-income fathers. | Inform practitioners about whether AID! Project design promotes healthy family relationships by improving parent behavior. |
| R2 | Low-income fathers can lack the <b>co-parenting skills</b> to fulfill their familial obligations as a parent to promote healthy family relationships. | Determine the extent to which the delivery of AID! Project services enhance the co-parenting skills of low-income fathers. | Inform practitioners about whether AID! Project design promotes healthy family relationships by improving co-parent behavior. |
| R3 | Low-income fathers can lack the <b>financial skills</b> to fulfill their familial obligations as managers of household finances to promote economic stability. | Determine the extent to which the delivery of AID! Project services enhance the financial management skills of low-income fathers. | Inform practitioners<br>about whether AID!<br>Project design<br>promotes economic<br>stability by improving<br>financial behavior. |
| R4 | Low-income fathers can lack parenting attitudes to facilitate the skills necessary to engage in healthy parenting behavior. | Determine the extent to which the delivery of AID! Project services enhance the <b>parenting</b> attitudes of low-income fathers. | Inform practitioners about whether AID! Project design promotes healthy family relationship by improving parenting attitudes. |

# 3. LOGIC MODEL

Clearly demonstrate how the research question(s) (and the related implementation features and/or participant outcomes) link to the proposed logic model and the theory of change for the program. You may append a copy of your logic model to this document.

Figure 1 in appendix A presents a logic model to specify a theory of change for delivering AID! *services*. Service delivery processes specified in the model are linked to the desired outcomes for healthy family relationships and economic stability. Model specification incorporates a Descriptive Study design to conceptualize service delivery to assess outcomes for the AID! Project by comparing primary and secondary participant outcomes before and after participants complete services.

<u>Service delivery processes</u>: Key aspects of service delivery processes in the theory of change—goals, inputs, activities, and outputs—articulate the experiences that are designed to solve specific problems for those who agree to participate in the AID! Project. As a result, three broad service delivery goals are identified to maximize AID! Project participation benefits as explained below:

- Goal 1 Deliver core curricula as primary services to AID! participants: Candidates will understand that they receive core curricula to develop their skills to engage in healthy behaviors for parenting, co-parenting, partner relations, employment, and financial management but only after receiving an orientation about the AID! Project and giving project staff informed consent to participate in study activities. Then, Father Factor, The Next Playbook, and Money Smart curricula will be delivered to participants as specified in the logic model.
- Goal 2 Deliver employment support services to AID! participants: Candidates will
  understand that they receive employment support services to develop their skills to engage
  in healthy behaviors for parenting, co-parenting, partner relations, employment, and
  financial management, but only after receiving an orientation about the AID! Project and
  giving project staff informed consent to participate in study activities. Then, Case Managers
  will help Job Coaches promote Job Readiness and help the Career Development Manager
  with job placement and post-employment success for participants.
- Goal 3 Conduct Continuous Quality Improvement (CQI) to ensure full implementation of primary and enhanced employment services to participants:
  Reports prepared and presented to the CQI Team by evaluators in each of the 5 steps in the CQI Process will use a series of performance indicators to track key outputs over time to identify any AID! services delivered that might fall short of the intended amounts to be offered (i.e., fidelity standards) and received (i.e., dosage thresholds) by them. The CQI Team will then work with project staff to develop and implement performance interventions to address any outputs that need improvement to ensure the services offered to and received by participants meet the intended amounts by the end of each program year.

<u>Desired Outcomes</u>: Outcomes specified in the logic model theorize the primary and secondary outcomes that are desired for participants after they complete *AID! services*. Secondary outcomes are the improved attitudes and expectations that indicate and reflect participant engagement in healthy parenting, partner relations, employment, and financial behaviors. Primary outcomes are the healthier behaviors exhibited by participants for parent, co-parent, and partner relationships that ultimately define the participation benefits for the AID! Project. All outcomes specified in the logic model are theorized to be more positive for eligible low-income fathers after they complete *primary services* and *post-employment support services*.

## 4. HYPOTHESES

For each specified research question, state the hypothesized result(s) and briefly describe why these results are anticipated.

| Research<br>Question | Hypothesized Result |
|---|---|
| R1 | Participants will report <b>healthier parenting behavior</b> one-year after they complete <i>primary services</i> and <i>employment support services</i> in the AID! Project. |
| R2 | Participants will report <b>healthier co-parenting behavior</b> one-year after they complete <i>primary services</i> and <i>employment support services</i> in the AID! Project. |
| R3 | Participants will report <b>healthier financial behavior</b> one-year after they complete <i>primary services</i> and <i>employment support services</i> in the AID! Project. |
| R4 | Participants will report <b>healthier parenting attitudes</b> immediately after they complete <i>primary services</i> and <i>employment support services</i> in the AID! Project. |

<sup>\*</sup> you may add rows by hitting the tab button, or right click and select insert row below

# 5. RESEARCH DESIGN

For each research question, briefly describe why the research design proposed will answer each research question(s). State whether the proposed evaluation is a <u>descriptive</u> or impact evaluation and justify why the proposed research design is best suited to answer the research question(s).

| Research Question | Design | Justification |
|---|---|---|
| R1 | Pre to follow-up assessment will estimate the impact of AID! participation on healthy parenting behavior. | Healthy change reported by participants in their parenting behavior from pre to 1-year follow-up estimates the maximum amount of benefit that can be attributed to AID! services in the absence of a counterfactual. |
| R2 | Pre to follow-up assessment will estimate the impact of AID! participation on healthy co-parenting behavior. | <b>Healthy</b> change reported by participants in their <b>co-parenting behavior</b> from pre to 1- <i>year</i> follow-up estimates the maximum amount of benefit that can be attributed to AID! services in the absence of a counterfactual. |
| R3 | Pre to follow-up assessment will estimate the impact of AID! participation on healthy financial behavior. | Healthy change reported by participants in their financial behavior from pre to 1-year follow-up estimates the maximum amount of benefit that can be attributed to AID! services in the absence of a counterfactual. |
| R4 | Pre to post assessment will estimate the impact of AID! | Healthy change reported by participants in their parenting attitudes from pre to post estimates the maximum amount of benefit that |

| participation | n on | healthy |
|---------------|--------|---------|
| parenting | attitu | udes. |

can be attributed to AID! services in the absence of a counterfactual.

## ONGOING GRANTEE AND LOCAL EVALUATOR COORDINATION

Describe how the grantee and local evaluator collaboratively worked together to identify the research question(s) and research design to ensure its feasibility and relevance. Describe how the grantee and local evaluator will continue to work together throughout the evaluation to proactively address unforeseen challenges as they arise and ensure the rigor and relevance of the evaluation and its findings. Describe how the grantee and local evaluator will coordinate dissemination efforts. Describe how these processes will occur while maintaining the independence of the evaluation.

The basis for ongoing coordination between Action for Children (the grantee) and MER (the local evaluator) is regular communication, by way of recurring meetings and daily interactions with embedded staff. Throughout the original proposal process, and now during the evaluation planning phase, MER worked in consort with AFC to design a study with research questions that are appropriate to the intervention. MER guides the process, given our experience designing and running evaluations, and AFC provides expertise on their community, target population, and program/curricula specifics.

Recurring meetings will include a bi-weekly project CQI team meeting. Under the leadership of the Data Manager and Lead MER Evaluator, the CQI team reviews data from the nFORM and local evaluation systems to identify and mitigate implementation or data issues, and closely examine trends and accomplishments. This team includes AFC organizational and project leadership, the MER Evaluation team, and front-line staff representatives (e.g., Facilitators, Case Managers).

In addition to CQI team meetings, overall project team meetings occur monthly (at a minimum), with project leaders across MER and AFC in attendance, to ensure the partnership remains strong and that coordination across organizations is on track. This recurring, ongoing meeting structure is conducive to close coordination, ensuring that challenges can be quickly addressed, and promising strategies can be efficiently maximized.

One of the key components of this coordination effort is the Data Manager, who is an AFC employee. The Data Manager functions to bridge the gap between organizations. They will interact with AFC staff daily while completing their job duties and play a leadership role in the recurring meetings outlined above. See Section II.D. above for more details about this role and others. Both the meetings and the roles outlined above will continue throughout the entire project period, providing opportunities to ensure the rigor and relevance of the evaluation and its findings, and to discuss and coordinate dissemination efforts (which will also be shared across MER and AFC).

MER has experience operating prior descriptive evaluations using this exact process. Clearly outlining roles and responsibilities maintains the independence of the evaluation. That is, the evaluation team helps identify and illuminate areas of concern or improvement (for the program and the evaluation), but the program staff have responsibility for implementing improvements and providing direct services to participants. In this way, AFC and MER acknowledge our shared interest in and responsibility for a well-executed project and evaluation, but that MER is also an

independent and external organization with a high level of integrity and is not responsible for nor invested in the specific outcomes of the program. This allows for close coordination without allowing for co-dependence, or for personal interests to influence evaluation findings.

## 7. LEAD STAFF

Define the roles of lead staff for the evaluation from both organizations below.

| Name | Organization | Role in the Evaluation |
|---|---|---|
| Dr. Matthew Shepherd | Midwest Evaluation and Research | Principal Investigator |
| Michelle Jackson, M.S. | Midwest Evaluation and Research | Evaluation Project Manager |

Articulate the experience, skills, and knowledge of the staff for the evaluation (including whether they have conducted similar studies in this field), as well as their ability to coordinate and support planning, implementation, and analysis related to a comprehensive evaluation plan.

Dr. Matthew Shepherd will serve as the Principal Investigator for this grant. As such, he has corporate responsibility for all evaluation activities. Dr. Shepherd has over 25 years' experience in program design and implementation, applied research, program evaluation, policy analysis, and evaluative technical assistance.

Michelle Jackson will serve as the Evaluation Project Manager. The Evaluation PM leads the effort to conduct a descriptive study <u>and</u> a Continuous Quality Improvement (CQI) process for the grant. Previously, Ms. Jackson has served as project lead for community foundation and grant evaluation projects. She has facilitated the data collection and survey tracking process for research assistants. In addition, she manages Midwest Evaluation's Institutional Review Board (IRB) submissions and reporting. In 2019, she was selected by Public Strategies as an Emerging Scholar to attend the 2019 Biennial Grantee Conference.

The CQI Data Manager will work closely with the grantee and community partners on-site to complete data collection and management activities for the descriptive study <u>and</u> a Continuous Quality Improvement (CQI) process.

#### 8. SAMPLE

# 8.1. TARGET POPULATION(S)

For each target population identified in Section 1.2, please describe the target population(s), and explicitly state whether the population(s) differs from those who will be broadly served by the grant. Describe how the target population will be identified. Explicitly state the unit of analysis (e.g., non-residential father, unmarried couple).

| Description of Target Population | How is the population different from those who will be broadly served by the grant? | How will the target population be identified? | Unit of<br>Analysis |
|---|---|---|---|
| 18+ year old urban<br>fathers in Franklin<br>County (OH) with<br>children age 24 and<br>under | No difference: all program participants will be study participants | The sample will be identified and recruited by the program staff. | Urban adult fathers |

# 8.2. POWER ANALYSIS

For each confirmatory outcome, please provide power analyses demonstrating proposed sample sizes will be able to detect expected effect sizes for the outcomes targeted. Refer to previous studies of similar interventions for estimates of the required sample to inform power analyses. Note: If an impact evaluation is not proposed, this issue does not need to be addressed. You may use the table below to report the assumptions used in your power calculations, as well as the resulting minimum detectable impact for your confirmatory outcomes or provide them in the space below.

Though not an RCT, the Power Analysis is as follows:

| | Outcome 1: | Outcome 2: | Outcome 3: |
|---|---|---|---|
| Outcome Name | Parenting Attitudes | Father<br>Relationship<br>Behavior<br>(parenting/co-<br>parenting) | Father Financial<br>Behavior |
| Continuous or binary? | Continuous | Continuous | Continuous |

| Level of significance (e.g., 0.05 percent) | 0.05 | 0.05 | 0.05 |
|---|---|---|---|
| Number of sides of test (one- or two-tailed) | 2 tailed | 2-tailed | 2-tailed |
| Power (e.g., 80 percent) | 80% | 80% | 80% |
| Total number of individuals in analytic sample | 483 | 483 | 483 |
| If continuous outcome, enter the standard deviation of the outcome (>0) | nFORM | nFORM | nFORM |
| Proportion of individual-<br>level (or within-group)<br>variance explained by<br>covariates | nFORM | nFORM | nFORM |
| Minimum detectable effect size | 0.030 | 0.030 | 0.030 |

# 8.3. METHODS TO PROMOTE SUFFICIENT PROGRAM PARTICIPATION

Please describe methods to promote sufficient program participation in the table below.

| What methods will you use to ensure sufficient sample is recruited, enrolls, and participates in the program? | Action for Children will over-recruit to ensure sufficient sample size. Incentives will be offered at various times in the curriculum to keep participants active. |
|---|---|
| Who will be responsible for recruiting the evaluation sample? | Applicants will be enrolled via street outreach or referral. Action for Children will use multiple targeted marketing platforms-such as billboards, radio, print, social media, flyers, brochures, and posters. Action for Children will also have an experienced and trained full-time recruiter, part-time recruiter, and other staff to assist in recruitment. |

Please describe any incentives to be offered for program participation and/or completion and/or data collection and/or participation in the evaluation.

Participants will be incentivized throughout participation in primary workshops as well for completing the one-year follow-up survey for evaluation purposes.

- \$25 gift card after completing Enrollment Surveys and attending 3 sessions
- \$25 gift card after the completion of Session 6
- \$75 gift card after the completion of Session 11 or 12 and the nFORM Post-Program Survey (& OLLE Post-Survey-only during evaluation enrollment period: ended 4/12/2024) if attendance is at least 90% for the core curriculum workshops

A \$50 gift card will be given for completion of the 1 Year Follow-Up Survey for evaluation purposes.

## 9. DATA COLLECTION

## 9.1. CONSTRUCTS AND MEASURES

Clearly articulate the constructs of interest, measures to evaluate those constructs, and specific data collection instruments. Provide any information on the reliability and validity of the data collection instruments. For standardized instruments, you may provide the citation for the instrument.

| Construct | Measure | Instrument | Reliability and Validity (if standardized instrument, you provide a citation for the instrument) |
|---|---|---|---|
| Parenting<br>Behavior<br>(interaction<br>with children) | 1 item: hours<br>spent w/children<br>in last 30 days<br>(interval); 1 item:<br>frequency reach<br>out to children<br>(categories, 5-<br>point scale); 7<br>items: frequency<br>engage in key<br>behaviors<br>(categories, 5-<br>point scale) | nFORM Community- Based Fathers Survey (A2b, A2c, A5b: b-d, f-i) *also asked on OLLE; will use data from survey with the most complete data | n/a |

| Co-Parenting<br>Behavior | 11 items:<br>frequency of<br>agreement with<br>key co-parenting<br>behaviors<br>(interval, 5-point<br>scale) | nFORM Community- Based Fathers Survey (A13: a-k) *also asked on OLLE; will use data from survey with the most complete data | n/a |
|---|---|---|---|
| Father Financial<br>Behavior | 2 items: yes or no<br>questions for<br>have resume,<br>checking/savings<br>accounts<br>(dichotomous) | nFORM<br>Community-<br>Based Fathers<br>Survey<br>(B3, B3a)<br>*also asked on<br>OLLE; will use<br>data from<br>survey with the<br>most complete<br>data | n/a |
| Parenting<br>Attitudes<br>(toward<br>children) | 7 items:<br>frequency of key<br>attitudes<br>(categories, 5-<br>point scale) | nFORM<br>Community-<br>Based Fathers<br>Survey (A3: a-g)<br>*also asked on<br>OLLE; will use<br>data from<br>survey with the<br>most complete<br>data | n/a |

# 9.2. CONSENT

Describe how and when program applicants will be informed of the study and will have the option of agreeing (i.e., consenting to) or declining to participate in the study.

Fathers will be recruited or referred to *All in Dads!*. Case Managers will contact fathers to fully explain the project, including the research component involving surveys at the start of workshops, the end of workshops, and 12-months following enrollment into the project. General intake information and the nFORM Applicant Characteristics Survey will be administered. At that point, an nFORM profile will be created. If the applicant decides to enroll in the project, the Case Manager will schedule the father for a virtual orientation session. If the applicant decides not to enroll in the project, he will be provided with resources and referrals to other programs. From there, fathers will attend their scheduled virtual orientation with a workshop facilitator where they will be reminded that participation in the project is voluntary, that they can drop out of the project at any time for any reason without consequences after completing the consent form and will be given the opportunity to leave the orientation session if they desire. If the applicant agrees to participate in the project, he will complete a consent form along with a release of information form, media release form, and the nFORM Entrance Survey. Informed consent will take place prior to program enrollment and the collection of evaluation data.

#### 9.3. METHODS OF DATA COLLECTION

If the evaluation will collect multiple waves of data, describe the timing of these waves below. When describing follow-up periods, specify whether the follow-up period will be post-baseline, post-random assignment, or post-program completion.

| Wave of Data Collection (e.g., baseline, short-term follow-up, long-term follow-up) | Timing of Data Collection |
|---|---|
| T1: baseline/pre-participation | Before first workshop session, at the same time as the nFORM entrance survey-following informed consent |
| T2: post-participation | After the final workshop session, at the same time as the nFORM exit survey |
| T3: 1-year follow-up | Collected approximately one year after program enrollment/baseline |

For each measure, describe how data will be collected detailing which data collection measures will be collected by which persons, and at what point in the programming or at what follow-up point.

| Measure | Timing of Data<br>Collection<br>(baseline, wave<br>of data<br>collection) | Method of Data<br>Collection | Who Is<br>Responsible<br>for Data<br>Collection? | Impact Evaluations Only: Will Methods or Collection Procedures Differ by Study Group? | Administrative Data Only: Will data access require data sharing agreement? |
|---|---|---|---|---|---|
| Parenting Behavior (interaction with children) 1 item: hours spent w/children in last 30 days (interval); 1 item: frequency reach out to children (categories, 5- point scale); 7 items: frequency engage in key behaviors (categories, 5- point scale) | nFORM Community Fathers Entrance Survey- administered at first workshop session/OLLE Pre; nFORM Community Fathers Exit Survey- administered at last workshop session/OLLE Post/OLLE Follow-Up | nFORM and/or OLLE Participant self-enters survey using online data collection platform | Case Manager/Facilita tor will proctor data collection and assist participants as necessary | | |
| Co-Parenting Behavior 11 items: frequency of agreement with key co-parenting behaviors (interval, 5-point scale) | nFORM Community Fathers Entrance Survey- administered at first workshop session/OLLE Pre nFORM Community Fathers Exit Survey- administered at last workshop session/OLLE Post/OLLE Follow-Up | nFORM and/or OLLE Participant self-enters survey using online data collection platform | Case Manager/Facilita tor will proctor data collection and assist participants as necessary | | |
| Father Financial<br>Behavior | nFORM<br>Community | nFORM and/or<br>OLLE | Case<br>Manager/Facilita | | |

| 2 items: yes or no<br>questions for have<br>resume,<br>checking/savings<br>accounts<br>(dichotomous) | Fathers Entrance Survey- administered at first workshop session/OLLE Pre; nFORM Community Fathers Exit Survey- administered at last workshop session/OLLE Post/OLLE- Follow-Up | Participant self-<br>enters survey<br>using online<br>data collection<br>platform | tor will proctor<br>data collection<br>and assist<br>participants as<br>necessary |
|---|---|---|---|
| Parenting Attitudes (toward children): 7 items: frequency of key attitudes (categories, 5- point scale) | nFORM Community Fathers Entrance Survey- administered at first workshop session/OLLE Pre; nFORM Community Fathers Exit Survey- administered at last workshop session/OLLE Post | nFORM and/or OLLE Participant self-enters survey using online data collection platform | Case Manager/Facilita tor will proctor data collection and assist participants as necessary |

# 9.4. ENSURING AND MONITORING DATA COLLECTION

Describe plans for training data collectors and for updating or retraining data collectors about procedures. Detail plans to regularly review data that have been submitted and to assess and swiftly address problems.

This evaluation will utilize both post-program surveys (completed at the completion of core programing) and follow-up surveys collected one year after enrollment / baseline. The methods for these data collections differ. The primary driver for post-program survey completion is high rates of program retention. This data point will be collected during the last workshop session – after (but during the same session of) the completion of the nFORM post-program data collection. As such only those individuals who complete the program and who are at the data collection session will participate in the post-program data collection.

All program staff and evaluation staff will undergo a rigorous set of trainings to prepare for the evaluation. All staff receive an overview and introductory training to present the goals and objectives of the evaluation effort and its importance to the overall project. Next all staff receive training on human subject's protection and are required to pass a certification test on the subject matter. All staff will also receive a detailed training on the details of the evaluation including the evaluation tools, timing and data collection process.

In addition, the Data Manager and the primary local evaluation staff will undergo a rigorous training process to better understand the context of HMRF research, training on data collection procedures they will be responsible for, and training on the nFORM system and use of nFORM data in a CQI process. MER is creating networks of CQI Data Managers and Evaluation Project Managers across the 12 projects that we are evaluating so that all staff have access to experienced Data Managers and evaluation staff who have done this work previously. This training takes the form of weekly training sessions that are currently under way.

Members of the CQI team will also receive specific training on the MER CQI process that has been developed prior to the launch of data collection or program services. As described elsewhere MER is assisting the program staff in implementing a robust CQI process that will focus on retention as one of the primary areas of program improvement and as such we are anticipating relatively modest levels of attrition for this data collection.

On a bi-weekly basis the Data Manager, the local evaluation staff and MER technical specialists will be responsible for downloading data from the nFORM and MER On-Line Local Evaluation (OLLE) systems for processing and presentation to the CQI team for tracking and monitoring performance measurement outcomes (recruitment, enrollment, dosage, completion, referrals, etc.) so that near real-time adjustments can be made to program implementation to ensure compliance with program goals and objectives.

All MER training is currently being recorded and as new staff come on board with projects or project staff turnover (or need refresher training), recorded training material can be shared and accessed with follow-up one on one training with the primary local evaluator and the MER Line of Business Lead.

## 9.5. TRACKING PARTICIPANTS AND REDUCING ATTRITION

If participants will complete post-program and/or follow-up surveys, please provide estimated response rates for each wave of data collection listed in 10.3. Please describe plans for tracking

participants and reducing attrition below. <u>Note: If no post-program or follow-up surveys are proposed, this issue does not need to be addressed.</u>

| For each wave of data |
|----------------------------|
| collection listed in 10.3, |
| what is your estimated |
| response rate? |

| Baseline | T1: 100%-done at time of enrollment/orientation |
|----------|-------------------------------------------------|
| Wave 1 | T2: 90%-Estimated completion rate |
| Wave 2 | T3: 70%-Estimated 1 year follow-up |
| Wave 3 | |
| Wave 4 | |

What steps will be taken to track participants to conduct follow-up surveys with as many participants as possible?

This evaluation will utilize both post-program surveys, administered after the completion of core programing, and follow-up surveys, collected one year after enrollment/baseline. The data collection methods for the two time periods will differ, and both have been successfully implemented by MER in prior studies.

The post-survey data point will be collected during the last workshop session, after the completion of the nFORM post-program data collection, so only those individuals who complete the program and who are at the data collection session will participate in the post-program data collection. Therefore, the primary driver for post-program survey completion is high rates of program retention. The grantee-evaluator joint CQI process will focus on retention as one of the primary areas of program improvement, and as such we are anticipating relatively modest levels of attrition for this data collection.

Tracking and data collection for the follow-up survey one year after baseline will be conducted differently, using an intent-to-treat model in which all participants enrolled are included in the follow-up survey data collection process. Participant tracking will begin at enrollment, where detailed tracking information will be collected during the informed consent process. This includes currently available traditional contact information for each participant (address, phone, email), as well as social media contact information (e.g., Facebook, Twitter), and detailed information for secondary contacts who will likely always be in contact with the participant (e.g., parents, siblings, friends). The consent form will obtain permission to contact these secondary sources to locate the participant for follow-up interviews, if necessary. Additionally,

\$50 Walmart gift cards are planned as incentives to encourage completion and show respect for the time of the participant.

Tracking will begin 60 days prior to the target survey due date, when a postcard that includes information about online or phone survey completion will be mailed to the provided contact address for the participant. The primary purpose of this postcard is to verify the address provided. When retuned mail is received because the participant no longer lives at the provided address, or the address is invalid, then the participant will be moved into a queue for tracking by MER trained research staff. If the postcard is not returned and the survey not completed, a formal letter will be mailed (and emailed if possible) to the participant at 60 days prior to the due date, again containing information for survey completion. The postcard and letter may help ensure MER name recognition in the event research staff do need to contact a participant directly by phone.

At 30 days prior to the survey due date, the participant will receive a phone call from MER staff directly to compete the follow-up survey. MER staff will attempt to reach the client with the phone information provided and via social media. If the client is unable to be contacted after 3 attempts, MER staff move the participant into the queue for more structured tracking, including through secondary contacts, and an iterative process of outreach and tracking will take place until the survey is complete, or all tracking efforts are exhausted.

For participants moved into the queue for tracking, the following steps are followed. MER will begin tracking by outreach to secondary contacts, which includes sending a letter for the participants to the address for the secondary contact, sending a letter to the secondary contacts themselves, and attempting to call the secondary contacts to get updated contact information for the participants. It should be noted that secondary contacts are never told details of the program the participants are in, or details that could violate confidentiality. Tracking may also include utilizing publicly available databases and services which MER has subscriptions for to obtain new or unknown contact information.

Please describe a plan for monitoring both overall and differential attrition (across treatment and comparison groups).

Overall attrition will be mitigated through the use of incentives granted to participants at upon completion of:

- Session 3 and complete entrance surveys
- Session 6
- Session 12 and complete the exit surveys
- 1 Year Follow-Up Survey

## 10.PRIVACY

Specify how the methods for data collection, storage, and transfer (e.g., to the federal government) will ensure privacy for study participants.

For these evaluation efforts Action for Children and MER will utilize nFORM for performance measurement data collection and storage, Qualtrics Enterprise for the collection and storage of local evaluation (OLLE) data, and Dropbox Enterprise for the storage of all data exported from either data collection system and all other program and evaluation documents. Logins with secure passwords will be necessary for all staff to access data they are authorized to enter/view. Using SPSS as our preferred statistical analysis and data management program, the highly experienced MER staff can combine and link data from multiple sources (including nFORM, Qualtrics, and other administrative data systems) into a complete data set with relative ease.

## nFORM

The nFORM system is a management information system that each HMRF grantee will use to collect and store the information that will be reported to the Office of Family Assistance (OFA) within ACF. The data from nFORM can also be easily exported to other programs, such as Microsoft Excel. The nFORM data will be entered by participants directly and by program staff (Case Managers, Facilitators, Project Director, and Data Manager) and the Data Manager will have the primary responsibility for overseeing the completeness, accuracy, and timeliness of data entered by staff. MER evaluation staff will download and analyze this data on a bi-weekly basis. nFORM will capture performance management data (including program operations, services, and client characteristics).

# **Qualtrics Enterprise**

Qualtrics is an industry leader in data collection and security and will be used for the collection and storage of participant responses to surveys for the local evaluation effort. This data will be entered directly by participants and by MER evaluation staff. Participants will use a provided link on tablets, computers, or phones to directly answer survey questions. Information collected in Qualtrics will be about outcomes, life situation, and other status indicators.

Qualtrics servers are protected by high-end firewall systems and scans are performed regularly to ensure that any vulnerabilities are quickly found and patched. Application penetration tests are performed annually by an independent third-party. All services have quick failover points and redundant hardware, with backups performed daily. Access to systems is restricted to specific individuals who have a need-to-know such information and who are bound by confidentiality obligations. Access is monitored and audited for compliance.

Qualtrics uses Transport Layer Security (TLS) encryption (also known as HTTPS) for all transmitted data. Surveys may be protected with passwords. Our services are hosted by trusted data centers

that are independently audited using the industry standard SSAE-18 method. Qualtrics has ISO 27001, FedRAMP and HITRUST authorization and certification. Information is easily and securely downloadable at any time to Excel or comma-separated formats and data in transit is secured using secure TLS cryptographic protocols. Qualtrics data is also encrypted at rest.

## **Dropbox**

Once data is downloaded by MER it is at all times stored on cloud-based storage provided by Dropbox Enterprise. All MER staff are prohibited from storing any project information (including data) on local computer hard drives. This ensures safety of the data from loss or unauthorized access due to the damage or theft of computers.

Dropbox adheres to the most stringent compliance standards by combining major accepted standards with compliance risk assessment measures, including ISO 27001, SOC 1, 2, and 3, GDPR, the CSA Code of Conduct, and HIPAA/HITECH. Data is also protected from data security threats with in-transit and at-rest encryption. The Dropbox Enterprise system also allows MER to recover accidentally deleted content and undo unwanted file changes, for up to 10 years. The Advanced Team & Content Controls Add-On, powered by BetterCloud technology, allows IT admins to deploy Dropbox on team devices and govern data in one place.

## 11.IRB/PROTECTION OF HUMAN SUBJECTS

Please describe the process for protection of human subjects, and IRB review and approval of the proposed program and evaluation plans. Name the specific IRB to which you expect to apply.

Because the planned evaluation involves human subjects, AFC understands that program implementation requires both IRB approval and participant informed consent. MER has an established relationship with Solutions IRB. MER has had 14 research studies approved by Solutions IRB over the past four years, completed over 15 annual check-in reports, and has submitted timely amendments when changes to studies needed to take effect. Solutions IRB, a private commercial Association for the Accreditation of Human Research Protection Programs Inc. (AAHRPP) fully accredited Institutional Review Board, will ensure that this study is approved before any research activities take place.

All submissions are completed online, so turnaround for a new study approval is between 24 to 72 hours, though the full approval process can take approximately one to two weeks depending on the number of questions and requested revisions that the IRB makes. In the IRB application submission, we will include descriptions of project staff, locations of study sites, the funding source, incentives, summary of activities, participant population, recruitment plans, risks and benefits, confidentiality of data, and the informed consent process along with all materials to be used in the study such as participant forms and surveys.

This project will be submitted for IRB approval in early March during the planning period in order to receive official approval to begin enrollment and data collection beginning in April.

Program staff and facilitators will also obtain Human Subjects Training Certification through the IRB to ensure the protection of participants.

## 12.DATA

#### 12.1. DATABASES

For each database used to enter data, please describe the database into which data will be entered (i.e., nFORM and/or other databases), including both performance measure data you plan to use in your local evaluation and any additional local evaluation data. Describe the process for data entry (i.e., who will enter the data into the database).

| Database Name | Data Entered | Process for Data Entry |
|---|---|---|
| nFORM | Performance Measurement<br>Data | Entered directly by participants, and by program staff |
| Qualtrics | Local evaluation data, participant outcomes (OLLE surveys) | Entered directly by participants, and by MER evaluation staff |

<sup>\*</sup> you may add rows by hitting the tab button, or right click and select insert row below

## 12.2. DATA REPORTING AND TRANSFER

For each database provided in the table above, please indicate the ability to export individual-level reports to an Excel or comma-delimited format and whether identifying information is available for linking to data from other sources.

| Database Name | Ability to Export Individual Reports? | What identifying information is available to facilitate linking to other data sources? |
|---|---|---|
| nFORM | capabilities of nFORM 2.0 unknown at this time | capabilities of nFORM 2.0 unknown at this time |
| Qualtrics | Yes, Excel or comma separated | Name, date of birth, gender, address, email, phone number |

## 12.3. CURRENT SECURITY AND CONFIDENTIALITY STANDARDS

For each database provided in Section 11.1, please Indicate the ability to be able to encrypt data access during transit (for example, accessed through an HTTPS connection); be able to encrypt data at rest (that is, when not in transit), have in place a data backup and recovery plan; require all users to have logins and passwords to access the data they are authorized to view; and have current anti- virus software installed to detect and address malware, such as viruses and worms.

| Database Name Ability encryp | Ability to encrypt at rest? | Backup and | Require all users to have logins | Current Anti-<br>Virus Software<br>Installed? |
|---|---|---|---|---|
|---|---|---|---|---|

| | data during transit? | | Recovery Plan? | and passwords? | |
|---|---|---|---|---|---|
| nFORM | Yes | Yes | Yes | Yes | Yes |
| Qualtrics | Yes | Yes | Yes | Yes | Yes |

| | (target population | is urban fathers who are 18+ years with child | ren up to 24 years who are residents of | Frankli | in County in Ohio) | | |
|---|---|---|---|---|---|---|---|
| Service delivery processes: | | | | | Desired outcomes: | | |
| 5 weeks duration for primary services and one year for CQI | | | | | assessed at enrollment and 1 year later | | |
| Goals: Increase participant capacity to promote healthy family relationships and economic stability. Inputs: Make the investments to deliver the intended service amounts to participants. | | <u>Activities</u> : Take the steps to ensure participants are offered and receive the intended service amounts. | <u>Outputs</u> : Track <i>quantifiable results</i> from activities to ensure service outputs meet standards and thresholds for participant offerings and dosage. | | Secondary: improved attitudes<br>and expectations indicative of<br>healthy family relationship and<br>economic stability behaviors. | | <u>Primary</u> : improved<br>behaviors for healthy<br>family relationships and<br>economic stability. |
| Goal 1: Deliver core curricula as p | rimary services to participants | s (n = 990 (90 in yr 1, 180 in yr 5) + (240 in yrs 2-4)). | | | | | |
| skills to engage in healthy parenting, co-parenting, partner relationship, and financial behaviors. Evidence-based curricu (Father Factor, The Ne Playbook, Money Sma Trained facilitators; Cla | Primary (core curricula):<br>Evidence-based curricula<br>(Father Factor , The New<br>Playbook , Money Smart ); | Father Factor (16 hrs = eight 2-hour sessions): Skills-based education to promote healthy parent, coparent, and partner relationships. The New Playbook (4 hrs = eight half-hour sessions): | Participants offered (990) and receive (594) 16 hours of <i>Father Factor</i> curricula (60% complete). | | Participants report | | |
| | Trained facilitators; Class space; Virtual meeting platforms | Skills-based education to promote healthy attitudes and behaviors to address violence and toxic masculinity. | Participants offered (990) and receive (594) 4 hours of <i>The New Playbook</i> curricula (60% complete). | | | | Participants repor |
| | | Money Smart (4 hrs = 2 two-hour sessions): Skills-based education to promote sound money management, budgeting, and credit building and repairing. | Participants offered (990) and receive (594) 4 hours of <i>Money Smart</i> (60% complete). | | improved attitudes and expectations (pre to | \ | engaging more<br>frequently in<br>healthy behaviors |
| Goal 2: Deliver employment suppo | ort services to participants (n | = 990 (90 in yr 1, 180 in yr 5) + (240 in yrs 2-4)). | | | post) that facilitate | | (pre to post) for |
| Problem: Many fathers may need<br>support to increase the<br>likelihood they will participate in<br>and benefit from primary | Managers, Job Coaches, | and remove barriers (job uniforms, bus passes, child care referrals). | pe job access (soft job skills training, related services) Participants offered (up to 990) and receive (up prove barriers (job uniforms, bus passes, child care ls). Participants offered (up to 990) and receive (up prove (up | | healthy behaviors for<br>family relationships<br>(parent, co-parent,<br>partner) and economic | 7 | family<br>relationships<br>(parent, co-parent |
| I ' | platforms (i.e. Zoom, Google<br>Meet, Microsoft Teams) | Post-Employment Support (Case Manager, Career Deve<br>Follow up with employment, internship, and apprenticeship<br>partners to ensure a successful transition for participants<br>and maintain relationships. | Participants offered (up to 990) and receive (up to 594) on-going Post-Employment (complete). | | stability. | , | partner) and<br>economic stability |
| Goal 3: Conduct Continuous Quali | ty Improvement (CQI) to ensu | re full implementation of project services. | | | | | |
| participants must be improved to | collection systems and carry | CQI Team (ongoing bi-weekly meetings): CQI Team uses a 5-step process to develop interventions that improve performance trends for service output indicators. | CQI team implements intervention strategies and assesses their impact on performance trends for service output indicators and outcomes (complete schedule CQI Reports for Steps 4-5). | | | | |

#### CONSORT Diagram for Action For Children: All In Dads!- Descriptive Evaluation

Eligible individuals are low-income urban fathers (custodial and noncustodial) in high poverty, high risk neighborhoods in Franklin County (OH), age 18 and above with children under 24 years of age.

Informed consent is obtained after the study is explained to interested potential participants. The target for program recruitment is 1080 people, to ensure 90 study participants in Year 1, 240 study participants in Year 2, 240 in Year 3, 240 in Year 4, and 180 in Year 5.

Study enrollment will end 3/31/24. No participants will be enrolled into the study for year 5 to allow time to collect the 1-year follow-up survey. Breakdown for study enrollment: year 1: 90, year 2: 240, year 3: 240, year 4: 120 equaling 690. Study Enrollment Period: 4/1/21 – 3/31/2024

Program Enrollment Period: 4/4/21-9/30/25

Evaluation Surveys Administered: 4/1/21 – 3/31/24

